CLINICAL TRIAL: NCT05793099
Title: Effect of 5% Aqueous Propolis Added to Sugar-Free Chewing Gum in Salivary and Dental Plaque pH in Children (in Vivo Study)
Brief Title: Effect of 5% Aqueous Propolis in Salivary and Dental Plaque pH in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UDDS-Pedo-05-2023
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Child; Saliva; Dental Plaque
Keywords: Aqueous Propolis; Chewing gum
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aqueous propolis 5% gum (Experimental): The children will be given aqueous propolis gums to chew for 15 minutes.
  Interventions: Other: Effect of aqueous propolis gums in salivary and dental plaque pH in children
- Placebo gum (Placebo Comparator): The children will be given placebo gums gums to chew for 15 minutes.
  Interventions: Other: Effect of placebo gums in salivary and dental plaque pH in children

INTERVENTIONS:
Other: Effect of aqueous propolis gums in salivary and dental plaque pH in children — The child will be given a 10% sucrose solution, and the salivary pH will be measured before and after giving sucrose solution (Baseline) and then the child will be given aqueous propolis gum to chew for 15 minutes to stimulate salivation. The saliva pH will be measured by taking a sample of the patient's saliva (3ml) while chewing the gum in the mouth in a disposable container and then saliva pH will be measured.
  Dental plaque pH also will be measured before and after administration of a 10% sucrose solution (Baseline), and then 15 minutes after chewing aqueous propolis gum dental plaque will be collected using the "plaque collection" technique from the 6 buccal surfaces of teeth 16,21,26,36,41,46 using a sterile excavator. The sample will be mixed with 0.05 ml of distilled water until it dissolves and then dental plaque pH will be measured.
  Arms: Aqueous propolis 5% gum
Other: Effect of placebo gums in salivary and dental plaque pH in children — The child will be given a 10% sucrose solution, and the salivary pH will be measured before and after giving sucrose solution (Baseline) and then the child will be given placebo gum to chew for 15 minutes to stimulate salivation. The saliva pH will be measured by taking a sample of the patient's saliva (3ml) while chewing the gum in the mouth in a disposable container and then saliva pH will be measured.
  Dental plaque pH also will be measured before and after administration of a 10% sucrose solution (Baseline), and then 15 minutes after chewing placebo gum dental plaque will be collected using the "plaque collection" technique from the 6 buccal surfaces of teeth 16,21,26,36,41,46 using a sterile excavator. The sample will be mixed with 0.05 ml of distilled water until it dissolves and then dental plaque pH will be measured.
  Arms: Placebo gum

SUMMARY:
This study aims to investigate the changes in saliva and dental plaque pH after consuming sugar-free chewing gum containing 5% of aqueous propolis in children aged between 8-11 years. The studied sample will be divided into two groups: Group A (Control group) placebo chewing gum, and Group B (Experimental group) aqueous propolis chewing gum. All children will experience both types of chewing gum with an interval of 1 week between the two studied groups.

DETAILED DESCRIPTION:
This study will evaluate saliva and dental plaque pH after consuming 10% sucrose solution and then each child will test each of the two types of gum (aqueous propolis 5% and placebo gum) so that the child himself is the control and tested sample together, according to the following order:

* In the first visit: the pH of saliva and dental plaque will be measured (before giving the sucrose solution, while chewing one of the two types of gum, and after giving the sucrose solution).
* In the second visit: after a week, the pH of saliva and dental plaque will be measured (before giving the sucrose solution, while chewing the other types of gum, and after giving the sucrose solution).)

ELIGIBILITY:
Inclusion Criteria:

1. Children have mixed occlusion.
2. Integrity of the buccal surfaces of the reference teeth (16, 21, 26, 36, 41, 46) from caries and developmental disorders
3. Children with DMFS ≥5 according to WHO guidelines and standards.

Exclusion Criteria:

1. Systematic or mental disorders
2. Medications that may affect the salivary flow rate or composition.
3. Allergy to natural sugar substitutes.
4. Children who wear fixed or removable orthodontic appliances.
5. Children who have the habit of daily use of sugar substitute products.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Saliva pH measurement | 5 minutes after chewing gum.
  saliva pH will be measured by using saliva pH meter.
Saliva pH measurement | 10 minutes after chewing gum.
  saliva pH will be measured by using saliva pH meter.
Saliva pH measurement | 15 minutes after chewing gum.
  saliva pH will be measured by using saliva pH meter.

SECONDARY OUTCOMES:
Dental plaque pH measurement | 15 minutes after chewing gum.
  Dental plaque will be Orion SA 720 pH/ISE Meter

CONTACTS AND LOCATIONS:
Overall Officials: Iman J Alahmad, DDs, Principal Investigator — MSc student in Pedodontics, University of Damascus; Shadi Azzawi, Phd, Study Director — Professor of Pedodontics, Department of Pedodontics, University of Damascus
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar S, Sogi SH, Indushekar KR. Comparative evaluation of the effects of xylitol and sugar-free chewing gums on salivary and dental plaque pH in children. J Indian Soc Pedod Prev Dent. 2013 Oct-Dec;31(4):240-4. doi: 10.4103/0970-4388.121822. PMID 24262397
- [Background] Gargouri W, Kammoun R, Elleuche M, Tlili M, Kechaou N, Ghoul-Mazgar S. Effect of xylitol chewing gum enriched with propolis on dentin remineralization in vitro. Arch Oral Biol. 2020 Apr;112:104684. doi: 10.1016/j.archoralbio.2020.104684. Epub 2020 Feb 19. PMID 32120052
- [Background] Toors FA. [Chewing gum and dental health. Literature review]. Rev Belge Med Dent (1984). 1992;47(3):67-92. French. PMID 1305985
- [Background] Monteil J, Hadj-Sassi A, Dargelos E, Guzman-Barrera N, Poque E, Leal-Calderon F. Method to prepare aqueous propolis dispersions based on phase separation. Food Chem. 2022 Sep 30;389:133072. doi: 10.1016/j.foodchem.2022.133072. Epub 2022 Apr 25. PMID 35490523
- [Background] Abbasi AJ, Mohammadi F, Bayat M, Gema SM, Ghadirian H, Seifi H, Bayat H, Bahrami N. Applications of Propolis in Dentistry: A Review. Ethiop J Health Sci. 2018 Jul;28(4):505-512. doi: 10.4314/ejhs.v28i4.16. PMID 30607063